CLINICAL TRIAL: NCT02692014
Title: A Multicenter Retrospective Observational Study on Different Risk Factors in Coronary Artery Stenosis Progression of CHD in China
Brief Title: Risk Factors Promoting Coronary Plaque Progression In China
Acronym: RIPPER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zhang Qi, MD (Other)
Responsible Party: Sponsor-Investigator, Zhang Qi, MD, Chief doctor, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: RJH20160126
Record Dates: First submitted 2016-02-21; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- coronary heart disease: 2,400 patients who are diagnosed with CHD and have received more than 2 times of coronary angiography within 12-24 months.

SUMMARY:
Coronary drug-eluting stent (DES) has been launched in China for more than ten years. Although it effectively decreases the overall incidence of re-stenosis, DES cannot inhibit the progression of atherosclerosis plaque outside segments. It was shown that the progression rate of non-target atherosclerosis plaque for patients with DES implantation was 6-10%, which indicated that current secondary prevention for coronary heart disease (CHD) is far from the achievement of ideal conditions.

Atherosclerosis has many risk factors based on current CHD guidelines, among which the level of low-density lipoprotein (LDL) is the most concerned one. Large clinical studies on statins were performed in the world during the past 20 years. It was demonstrated in these studies that statins were significant to both primary and secondary preventions of CHD. What's more, the lower of LDL level is reached, the lower incidence of clinical cardiovascular events is achieved. However, cardiovascular events were still not avoidable especially for the secondary prevention of CHD even if the level of LDL was significantly controlled under the recommended range of guidelines by high dosage of statins.

It was shown in some recent studies that high loading dosage of statins may effectively control the progression of coronary plaque. However, multiple studies found it was hard to control the progression of all patients of coronary plaque due to individual difference.

Currently China Food and Drug Administration (CFDA) has not approved the loading dosage of all statins because of possible high safety issues and confusions about the appropriate application in Chinese patients, as well as economy burden to Chinese patients with high treatment cost. How to evaluate individual progression risk of coronary plaque and enhance risk factors control and the treatment of statins for necessary population, is currently an issue, which should be solved in the diagnosis and treatment of CHD.

The inhibition in the progression of atherosclerosis plaque is not absolutely dependent on the decrease of LDL. Large number of studies found other risk factors. For instance, diabetes and chronic kidney diseases may also be associated with the progression of plaque. However, the potential impact and control are still uncertain up to date.

Based on these background, we design a retrospective study, Risk Factors Promoting Coronary Plaque Progression In China (The RIPPER Study), to solve these issues.

DETAILED DESCRIPTION:
STUDY DESIGN This is a national multicenter retrospective study. Through reviewing angiography database in 20 CHD intervention centers of China. We will collect the data of 2400 patients with twice of coronary angiography as well as 12-24 months interval from Jun 2013 to Dec 2016. We will confirm the actual rate in the coronary plauqe progression of CHD patients in China as well as regression analysis to investigate the impact of different risk factors on the progression of coronary plaque, thus find the primary risk factors and rational strategy in secondary prevention. In this study, the included patients should not be replaced or withdrawal.

STUDY POPULATION 2,400 patients who are diagnosed with CHD and have received more than 2 times of coronary angiography within 12-24 months will be enrolled. If the number of angiography is more than 2 times. Patients who receive examination not in the same coronary intervention center will not be included.

STUDY DURATION It will take 12 months to collect data of 2,400 cases in 20 CHD intervention centers of China and following 9 months to compete QCA and risk factors analysis STUDY PROCESS The statistical analysis will include all the materials of cases. We will describe the basic history characteristics of patients, test parameters and the imaging characteristics of coronary angiography. Continuous variables will be described by number, mean, standard deviation (SD), median, minimum value and maximum value. Numeric variables with normal distribution will be described by mean and SD. Continuous variables will be compared by student test (normal distribution) and Wilcoxon rank sum test (skew distribution). Categorical variables (nominal variables/rank variables) will be described as frequency and percentage, which can be compared by Chi square test or Fisher exact test. Logistic multiple regression can be used to evaluate the risk factors of coronary disease progression in Chinese patients, among which the possible risk factors selection is based on clinical and statistical decision. Receiver operating characteristic(ROC) curve can be used to establish risk evaluation model of coronary disease progression and evaluate its value. The incomplete data will not be analyzed.

Data analysis will be processed by SPSS 13.0. All the analysis will be used the 2-side test or 2-side 95% confidence interval. There is statistical significance if 2-side P value is less than 0.05. This study will use descriptive analysis and finally report primary and secondary outcomes by graphics.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* more than 2 times of CAG in the same coronary intervention center
* within 12-24 months during Jun 2013 to Dec 2016

Exclusion Criteria:

* CABG history prior to the last record of CAG
* poor imaging quality of CAG
* not consistent with the requirements of QCA analysis
* mediated by other non-atherosclerosis factors such as arteritis
* pregnant
* other factors considered as not appropriate for inclusion by investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It will take 12 months to collect data of 2,400 cases in 20 CHD intervention centers of China and following 9 months to compete QCA and risk factors analysis.
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Actual)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Risk factors | 12 months
  Risk factors of the decreased diameter of in situ coronary stenosis (percentage) or vascular occlusion is analyzed by QCA

SECONDARY OUTCOMES:
The extent of decreased diameter of in situ coronary stenosis | 12 months
  analysed by QCA
The progression of coronary stenosis | 12 months
  observed by coronary angiography(CAG), defined as 20% increase of stenosis without intervention.
ISR | 12 months
  The incidence of in stent restenosis

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China